CLINICAL TRIAL: NCT01964690
Title: Lactate and Sepsis : What Dosage Use as Triage Tool in Emergency Department for Patients With Suspected Infection.
Brief Title: Lactate Use as Triage Tool in Sepsis : Veinous, Capillary or Arterial?
Status: Completed | Type: Observational
Sponsor: Hopital Saint Roch (Other)
Responsible Party: Principal Investigator, Contenti Julie, AFERSAU, Hopital Saint Roch
Other Study IDs: CAL2013; 2013-AO1293-42 (Other: ANSM)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-01

CONDITIONS: Sepsis
Keywords: Lactate; Sepsis; Capillary lactate; Venous lactate; Quick test
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Severe sepsis and septic shocks are increasingly codified. A biomarker as Lactate is very interesting to detect those situations. Usually, lactate used is arterial but results are often too slow to obtain if we want to respect Surviving Sepsis Campaign guidelines. Some analyzers (EKF diagnostics Lactate Scout*) can give results in 15 seconds.

We hypothesized that capillary lactate, easy to sample, tested with this analyzer may detect earlier those infections states and we want to find the most accurate site to detect severe sepsis (capillary, venous or arterial sample).

DETAILED DESCRIPTION:
Actually, patients presenting a sepsis with arterial lactate> 2 mmol.l-1 must be considered as criticals, and if lactate> 4 mmol.l-1 as septic shock. However, results are usually slow to obtain, especially if we want to respect the Surving Sepsis Campaign, which preconize antibiotic as soon as possible (first hour).

In admission room, arterial sample can't be easily done and usual results need more than 30 minutes. On the contrary, using analyzers like "EKF diagnostics Lactate Scout*" can give results faster with capillary blood (15 seconds). We will compare this results with both veinous and arterial lactate.

* For primary outcome, we will determine the most accurate value of capillary or veinous lactate that may be able to detect critical patient suspected of infection.
* for secondary outcomes, we will determine if quick capillary lactate test may replace arterial lactate in this indication and be able to predict mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* S.I.R.S : 2 or more criteria (fever > 38.3°C or hypothermia (core temperature < 36°C) heart rate > 90.min-1, tachypnea, altered mental status)
* Suspected infection

Exclusion Criteria:

* Arterial sample by laboratory reference method no available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected infection in emergency department (admission time)
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Lactate value | At admission in emergency department
  Determine the most accurate value of capillary or venous lactate that may be able to early detect patients with severe sepsis or septic shock, using quick test (EKF diagnostics Lactate scout*).

SECONDARY OUTCOMES:
Comparison values of capillary lactate and arterial lactate | 30 minutes after sampling
  Determine if capillary blood lactate may replace laboratory reference method (arterial lactate)
Mortality | Day 28 mortality
  Determine if capillary lactate value can be use as a mortality predictive tool

CONTACTS AND LOCATIONS:
Overall Officials: Contenti Julie, M.D, Principal Investigator — Association pour la Formation l'Enseignement et la Recherche du Service de l'Accueil des Urgences; Jacques Levraut, PD,MD, Study Director — CHU de Nice, France
Locations (1):
- Hopital Saint Roch, Nice, Alpes-maritimes, France

REFERENCES:
- [Derived] Contenti J, Corraze H, Lemoel F, Levraut J. Effectiveness of arterial, venous, and capillary blood lactate as a sepsis triage tool in ED patients. Am J Emerg Med. 2015 Feb;33(2):167-72. doi: 10.1016/j.ajem.2014.11.003. PMID 25432592